CLINICAL TRIAL: NCT06619951
Title: A Clinical Trial to Evaluate the Effects of Itraconazole or Rifampicin on the Pharmacokinetics of VC004 Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC004-106
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced or Metastatic Solid Tumor
Keywords: Healthy Volunteers
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: VC004 and itraconazole (Experimental)
  Interventions: Drug: VC004 and Itraconazole
- Group 2: VC004 and rifampicin (Experimental)
  Interventions: Drug: VC004 and rifampicin

INTERVENTIONS:
Drug: VC004 and Itraconazole — A single dose of VC004 was administered in the period 1. and a single dose of VC004 and Itraconazole coadministration in the period 2.
  Arms: Group 1: VC004 and itraconazole
Drug: VC004 and rifampicin — A single dose of VC004 was administered in the period 1. and a single dose of VC004 and rifampicin coadministration in the period 2.
  Arms: Group 2: VC004 and rifampicin

SUMMARY:
This study will adopt a Single-center, Single-arm, Open, Fixed Sequence design to Evaluate the Effects of Itraconazole or Rifampicin on the Pharmacokinetics of VC004 Capsules in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent before study, and fully understand the study content, process and possible adverse reactions;
* Able to complete the study in compliance with the protocol;
* Subject (including partner) is willing to voluntarily take effective contraceptive measures from screening through 6 months after the last dose of study drug;
* Male and female subjects between the ages of 18 and 45 years, inclusive;
* At least 50.0kg for male subjects, 45.0kg for female subjects, with a Body Mass Index between 19.0-26.0 kg/m2, inclusive;

Exclusion Criteria:

* More than 5 cigarettes per day on average within 3 months prior to screening;
* with A history of allergies, including medications, foods, mites, etc., or those known to be potentially allergic to drugs similar to the study drug, or those known to be allergic to itraconazole, rifampicin, or any excipients;
* History of drug and/or alcohol abuse (alcoholism defined as: drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); history of drug abuse or or have used drugs within the past five years;
* Donation or loss of a significant volume of blood (>400 mL) within 3 months prior to screening;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day1-Day16
  Maximum Observed Plasma Concentration (Cmax)
Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC） | Day1-Day16

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Affiliated to Southeast University, Nanjing, Jiangsu, China